CLINICAL TRIAL: NCT03577457
Title: The Interaction Between Oxytocin and Serotonin on the Social-reward Brain Networks and Decision Making
Brief Title: The Interaction Between Oxytocin and Serotonin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Benjamin Becker, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: SANP-2017-3-ATD
Record Dates: First submitted 2018-02-05; First posted 2018-07-05 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Healthy
Keywords: oxytocin; serotonin; social reward; decision making
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- male oxytocin and ATD group (Experimental): male subjects receiving oxytocin and ATD treatment
  Interventions: Drug: oxytocin nasal spray; Drug: ATD treatment
- male oxytocin and placebo group (Experimental): male subjects receiving oxytocin and ATD-placebo treatment
  Interventions: Drug: oxytocin nasal spray; Drug: oral placebo treatment (placebo-control for ATD)
- male placebo and ATD group (Experimental): male subjects receiving oxytocin placebo and ATD treatment
  Interventions: Drug: ATD treatment; Drug: intranasal placebo treatment (placebo-control for oxytocin)
- male placebo group (Placebo Comparator): male subjects receiving oxytocin placebo and ATD placebo treatment
  Interventions: Drug: intranasal placebo treatment (placebo-control for oxytocin); Drug: oral placebo treatment (placebo-control for ATD)

INTERVENTIONS:
Drug: oxytocin nasal spray — intranasal administration of oxytocin (24 IU)
  Arms: male oxytocin and ATD group; male oxytocin and placebo group
Drug: ATD treatment — oral administration of ATD (75.2g) (Acute Tryptophan Depletion)
  Arms: male oxytocin and ATD group; male placebo and ATD group
Drug: intranasal placebo treatment (placebo-control for oxytocin) — intranasal administration of placebo nasal spray
  Arms: male placebo and ATD group; male placebo group
Drug: oral placebo treatment (placebo-control for ATD) — oral administration of a tryptophan-balanced mixture (78.2g)
  Arms: male oxytocin and placebo group; male placebo group

SUMMARY:
The primary objective of this study is to identify any interaction between oxytocin and serotonin on neural and behavioral activity related to social reward and decision making by a double-blind, placebo-controlled, between-subject, pharmacological fMRI design

DETAILED DESCRIPTION:
Serotonin and oxytocin have been proved to play an important role in social reward processing and decision making in human. The aim of this study is to determine whether they interact in those essential human behaviors by a double-blind, placebo-controlled, between-subject, pharmacological fMRI design, in which 4 groups of healthy males will be administered with a random combination of nasal oxytocin (24 international units, IU) or placebo and acute tryptophan depletion (ATD, 75.2g) or placebo (a tryptophan-balanced mixture, 78.2g). The social-reward related neural activity and behavior will be assessed by a series of social reward task in and out of fMRI scanner and the decision making will be assessed by reversal learning task, ultimatum game (UG) and loss aversion task. The interaction between serotonin and oxytocin on brain networks will also be tested by resting state.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without past or current psychiatric or neurological disorders
* Right-handedness

Exclusion Criteria:

* History of head injury;
* Medical or psychiatric illness.
* High blood pressure, general cardio-vascular alterations
* History of drug or alcohol abuse or addiction.
* Allergy against medications or general strong allergies
* Sleep disorders.
* Visual or motor impairments

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-06-20 (Estimated); Study Completion 2019-07-20 (Estimated)

PRIMARY OUTCOMES:
Changes in brain neural activity during the social reward processing as assessed via fMRI | approximately 45 minutes after intranasal administration of oxytocin, or placebo, approximately 5.5h after administration of ATD, or placebo
  Whole brain and region of interest (ROI) regression analysis will be used to compare the neural activity of participants in response to social reward task in different treatment groups.
Changes in the resting state as assessed via fMRI | Time Frame: approximately 45 minutes after intranasal administration of oxytocin, or placebo, approximately 5.5h after administration of ATD, or placebo
  Resting state activity in the social reward related and decision making brain networks will be compared between the treatment groups

SECONDARY OUTCOMES:
Associations with Personalities of subjects | before 30mins ATD or placebo administration
  Personalities of subjects will be measured by a series of scales related to decision making and social reward, such as the Sensitivity to Punishment and Sensitivity to Reward Questionnaire (SPSRQ), which measures participants' sensitivity to reward and punishment. SPSRQ is a self-reported instrument that includes 48 yes/no questions divided into two subscales: Sensitivity to Reward (SR, 24 items, ranging from 0 (insensitive) to 24 (sensitive) to reward) and Sensitivity to Punishment (SP, 24 items, ranging from 0 (insensitive) to 24 (sensitive) to punishment). Associations between individual differences in personalities of subjects and differences in behaviors will be measured.
Behavioral performance in decision making task | approximately 4h after administration of ATD, or placebo, before nasal spray
  Behavioral performance in reversal learning task will be measured and compared between treatment groups.
Behavioral performance in social reward related task | approximately 105 minutes after intranasal administration of oxytocin, or placebo, approximately 6.5h after administration of ATD, or placebo
  Behavioral performance will be measured and compared between treatment groups

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Normal University, Beijing, China